CLINICAL TRIAL: NCT01380457
Title: A Comparative Bioavailability Study of Dronabinol Capsules 10 mg Under Fasting Conditions
Brief Title: Bioavailability Study of Dronabinol Capsules 10 mg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: BASi Clinical Research Unit (Unknown)
Responsible Party: Alfred Elvin/Director of Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 11885
Record Dates: First submitted 2011-06-16; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: To Determine Bioequivalence Under Fasting Conditions
Keywords: bioequivalence; dronabinol; fasting
MeSH Terms: conditions — Fasting | interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received the test formulated product manufactured by Pharmaceutics International, Inc. and marketed by Par Pharmaceutical, Inc. under fasting conditions
  Interventions: Drug: Dronabinol
- B (Active Comparator): Subjects received the reference listed drug manufactured by Banner Pharmacaps, Inc. and marketed by Unimed Pharmaceutical, Inc.
  Interventions: Drug: Marinol

INTERVENTIONS:
Drug: Dronabinol — Capsules, 10 mg, single dose, fasting conditions
  Other Names: Marinol
  Arms: A
Drug: Marinol — Capsules, 10 mg, single-dose, fasting conditions
  Other Names: Dronabinol
  Arms: B

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of Dronabinol 10 mg capsules verses Marinol.

DETAILED DESCRIPTION:
To compare the plasma levels of dronabinol (delta-9-tetrahydrocannabinol)and the principle active metabolite 11-OH-delta-9-tetrahydrocannabinol levels produced after administration of the test formulation with those produced after administration of a marketed reference product, under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 18 - 55 years of age
* Subjects must be within 18 to 29.9 kilograms/m2 per the BMI
* General good health as determined by medical history and physical examination within 30 days prior to the start of the study
* Blood chemistry, hematology, and urinalysis tests will be performed within 30 days prior to the start of the study
* No participation in an investigational drug study or donation of blood within 30 days prior to the start of the study
* At screening, subjects must have blood pressure and pulse rate within specified ranges
* No grapefruit juice or grapefruit-containing products for at least 72 hours prior to drug administration, each period. Subjects will be queried at check-in each period on consumption of grapefruit juice or grapefruit containing products. Results will be recorded and reported in the final report.
* No alcohol consumption for at least 24 hours prior to drug administration, each period
* No caffeine or xanthine consumption for 48 hours prior prior to drug administration, each period
* No prescription drugs (excluding hormonal contraceptives) within 14 days prior to drug administration, each period
* Subjects should refrain from taking OTC preparations, and/or nutritional supplements within 7 days prior to drug administration, each period. Subjects shall refrain from taking herbal remedies within 14 day prior to drug administration, and throughout the study periods
* Female subjects must not be pregnant or nursing; and must be surgically sterile; one year post-menopausal; or on hormonal contraceptive agents), a diaphragm or condom with spermicidal foam or jelly, or IUD for at least 3 months prior to drug administration and agree to use the same method of contraception for at least 1 month after the last drug administration
* Negative serum pregnancy test at screening and negative urine pregnancy test prior to drug administration, each period
* Negative HIV 1, hepatitis B surface antigen, an urine screen for drugs of abuse within 30 days prior to the start of the study

Exclusion Criteria:

* Disease or condition that could impact interpretation of study results or a condition which treatment would be contraindicated per currently approved product labeling
* Subjects had any of the following conditions:

  * used any prescription or OTC medication within 14 days of study initiation
  * a positive urine test for illicit drugs
  * participated in a clinical investigation within the past 30 days
  * had clinically significant allergies to drugs or foods, ot
  * any condition that might place them at increased risk of complications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2006-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence
  To conclude bioequivalence; 90% geometric confidence interval was contained within the limits 0.8 to 1.25.

CONTACTS AND LOCATIONS:
Overall Officials: Dilip K Guha-Ray, M.D., Principal Investigator — BASi Baltimore Clinical Research Unit
Locations (1):
- BASi, Baltimore, Maryland, United States